CLINICAL TRIAL: NCT03207516
Title: Impact of Bakery Products With Sourdough or Brewer's Yeast on Digestive Function: a Double Blind Randomised Study in Healthy Subjects
Brief Title: Sourdough Bakery Products and Digestive Function
Acronym: Digeribilità
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irccs Sdn (Other)
Collaborators: Federico II University (Other); Fresystem S.p.A. (Unknown)
Responsible Party: Principal Investigator, EMANUELE NICOLAI, Principal Investigator, Irccs Sdn
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1-14_Digeribilità
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Dyspepsia
Keywords: sourdough; leavening process; fermentation; brewer's yeast
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sourdough --> Brewer's Yeast (Active Comparator): Sourdough --> Brewer's Yeast
  1. administration of two 100 g croissants prepared with sourdough after an overnight fast.
  2. Magnetic Resonance (MR) Imaging analysis of gastric emptying, evaluation of postprandial gastrointestinal fermentation, croissant palatability, gastrointestinal symptoms and perceptions, and serum glucose levels at several time points.
  3. washout period: 7 days
  4. administration of two 100 g croissants prepared with brewer's yeast after an overnight fast.
  5. Magnetic Resonance (MR) Imaging analysis of gastric emptying, evaluation of postprandial gastrointestinal fermentation, croissant palatability, gastrointestinal symptoms and perceptions, and serum glucose levels at several time points.
  Interventions: Dietary Supplement: Sourdough --> Brewer's Yeast; Dietary Supplement: Brewer's Yeast --> Sourdough
- Brewer's Yeast --> Sourdough (Active Comparator): Brewer's Yeast --> Sourdough
  1. administration of two 100 g croissants prepared with brewer's yeast after an overnight fast.
  2. Magnetic Resonance (MR) Imaging analysis of gastric emptying, evaluation of postprandial gastrointestinal fermentation, croissant palatability, gastrointestinal symptoms and perceptions, and serum glucose levels at several time points.
  3. washout period: 7 days
  4. administration of two 100 g croissants prepared with sourdough after an overnight fast.
  5. Magnetic Resonance (MR) Imaging analysis of gastric emptying, evaluation of postprandial gastrointestinal fermentation, croissant palatability, gastrointestinal symptoms and perceptions, and serum glucose levels at several time points.
  Interventions: Dietary Supplement: Sourdough --> Brewer's Yeast; Dietary Supplement: Brewer's Yeast --> Sourdough

INTERVENTIONS:
Dietary Supplement: Sourdough --> Brewer's Yeast — Impact of bakery products with sourdough or brewer's yeast on digestive function
Dietary Supplement: Brewer's Yeast --> Sourdough — Impact of bakery products with sourdough or brewer's yeast on digestive function

SUMMARY:
In a double-blind, randomised crossover study, two sourdough croissants (SC) or two brewer's yeast croissants (BC) were served to 17 (9 F; Age range 18-40; BMI range 18-24 kg/m2) healthy subjects to evaluate the effects of their ingestion on postprandial gastrointestinal functions. Hydrogen breath test was performed to measure H2 production after SC and BC ingestion. Gastric volume was evaluated by Magnetic Resonance(MR) Imaging to calculate gastric emptying rate in the 3-hour interval following croissant ingestion. Palatability and postprandial gastrointestinal symptoms and perceptions over a 4-h period after the meal were evaluated by visual analogue scale (VAS). In addition, in the 3-hour interval, blood samples were drawn to measure serum glucose levels. The area under the curve (AUC) was employed to evaluate global kinetics of all parameters and the T-test was used to evaluate differences between groups.

DETAILED DESCRIPTION:
In this monocentric study, a double-blind, randomised crossover design was used, with washout periods of at least one week between study days. A standardized meal consisting of two 100 g croissants prepared with sourdough or with brewer's yeast was administered randomly to 17 (9 F; Age range 18-40; BMI range 18-24 kg/m2) healthy subjects after an overnight fast (at least 8 h) and consumed in a 10-minute interval with 300 mL of water. Immediately after meal ingestion, subjects were asked to evaluate croissant palatability. Gastric volume was evaluated by Magnetic Resonance(MR) Imaging to calculate gastric emptying rate in the 3-hour interval following croissant ingestion. Hydrogen breath test was performed to assess gastrointestinal fermentation measuring H2 production after SC and BC ingestion. Postprandial gastrointestinal symptoms and perceptions over a 4-h period after the meal were evaluated by visual analogue scale (VAS). In addition, in the 3-hour interval, blood samples were drawn to measure serum glucose levels. The protocol was repeated twice in each subject, once with sourdough croissants (SC) and once with brewer's yeast croissants (BC), dispensed according to a computer generated randomisation list created by RC following simple randomisation procedures (computerized random numbers). The area under the curve (AUC) was employed to evaluate global kinetics of all parameters and the T-test was used to evaluate differences between groups.

ELIGIBILITY:
Inclusion criteria:

* age ranging between 18 and 40 yrs
* normal-weight (body mass index 18-24.9 kg/m2),

Exclusion criteria:

* smoke
* functional or organic gastrointestinal disease
* gluten allergy
* dyslipidemia
* diabetes
* psychiatric disorders
* claustrophobia
* pregnancy
* breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2015-04-28 (Actual); Study Completion 2015-04-28 (Actual)

PRIMARY OUTCOMES:
Change of gastric emptying | 0, 3, 6, 9, 12, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180 minutes after the ingestion of the test meal
  Gastric volume in mL was evaluated by Magnetic Resonance(MR) Imaging using a 3-Tesla MR scanner (Biograph mMR, Siemens Healthcare, Erlangen, Germany) to calculate gastric emptying rate in the 3-hour interval following croissant ingestion

SECONDARY OUTCOMES:
Change of gastrointestinal fermentation | The hydrogen concentration in end expiratory air (expressed in ppm) was determined before consuming the test meal and then at 45, 60, 90, 120, 150, 180 and 240 minutes following meal ingestion.
  Hydrogen breath test (Gastrolyzer+TMMedimar) was performed to measure H2 production expressed in ppm after SC and BC ingestion
Palatability | Croissant palatability was evaluated immediately after meal ingestion
  Palatability were evaluated by visual analogue scale (VAS, expressed in mm)
Change of gastrointestinal symptoms | The presence and severity of gastrointestinal symptoms were assessed before test meal ingestion and at 45, 60, 90, 120, 150, 180 and 240 minutes after ingestion.
  postprandial gastrointestinal symptoms (gastrointestinal discomfort, bloating, nausea, fullness) were evaluated by visual analogue scale (VAS, expressed in mm) over a 4-h period after the meal
Change of gastrointestinal perceptions | The presence and severity of gastrointestinal perceptions were assessed before test meal ingestion and at 45, 60, 90, 120, 150, 180 and 240 minutes after ingestion.
  postprandial gastrointestinal perceptions (hunger, appetite, satiety and gastrointestinal wellbeing) were evaluated by visual analogue scale (VAS, expressed in mm) over a 4-h period after the meal
Glycemic profile | Blood samples were collected before test meal ingestion and at 15, 45, 60, 90, 120 and 180 minutes after the meal.
  blood samples were drawn to measure serum glucose levels in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Nicolai, Principal Investigator — Irccs Sdn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polese B, Nicolai E, Genovese D, Verlezza V, La Sala CN, Aiello M, Inglese M, Incoronato M, Sarnelli G, De Rosa T, Schiatti A, Mondelli F, Ercolini D, Cuomo R. Postprandial Gastrointestinal Function Differs after Acute Administration of Sourdough Compared with Brewer's Yeast Bakery Products in Healthy Adults. J Nutr. 2018 Feb 1;148(2):202-208. doi: 10.1093/jn/nxx049. PMID 29490103